CLINICAL TRIAL: NCT06216717
Title: Study of the Location of Motor Cortical Stimulation Electrodes in Chronic Neuropathic Refractory Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 24Neurochir01
Record Dates: First submitted 2024-01-11; First posted 2024-01-22 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Neuropathic Pain
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cortical stimulation has been used since 1991 to treat neuropathic pain. However, the underlying mechanisms are still incompletely understood and under-studied. In this protocol, the investigators aim to study the myeloarchitectonic and functional characteristics of areas activated by cortical epidural electrodes and to determine their relation to therapy response in chronic neuropathic refractory pain patients.

ELIGIBILITY:
Inclusion Criteria

* adults
* patient implanted with a motor cortical stimulation system for chronic neuropathic refractory pain,
* patient with available postoperative scanner

Exclusion Criteria: None

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: adults who were implanted with a motor cortical stimulation system for treatment of chronic neuropathic refractory pain between 2003-2023
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-01-20 (Estimated); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Pourcentage of pain relief | 1 year
  percentage of pain relief for different stimulated areas

SECONDARY OUTCOMES:
location of leads on the postoperative imaging | 1 month
  location of leads on the postoperative imaging

CONTACTS AND LOCATIONS:
Overall Officials: Petru ISAN, Principal Investigator — Centre Hospitalier Universitaire de Nice